CLINICAL TRIAL: NCT07336160
Title: Effect of ERAS-Based Preoperative Nutrition Education and Fasting Protocol on Postoperative Hydration Status and Nausea-Vomiting in Patients Undergoing Total Knee Arthroplasty
Brief Title: ERAS-Based Preoperative Nutrition and Fasting in Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nermin Ocaktan (Other)
Responsible Party: Sponsor-Investigator, Nermin Ocaktan, Assistant Professor, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12/474
Record Dates: First submitted 2025-12-26; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty; Postoperative Nausea and Vomiting
Keywords: Enhanced Recovery After Surgery; ERAS Protocol; Preoperative Nutrition; Fasting Protocol; Total Knee Replacement; Postoperative Hydration; Nausea and Vomiting; Perioperative Nursing Care
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups: an intervention group receiving ERAS-based preoperative nutrition education and fasting protocol, and a control group receiving standard care. Outcomes will be assessed preoperatively and postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS-Based Preoperative Nutrition and Fasting Protocol Group (Experimental): Participants receive ERAS-based preoperative nutrition education and an evidence-based fasting protocol during the 24 hours before total knee arthroplasty.
  Interventions: Behavioral: ERAS-Based Preoperative Nutrition Education and Fasting Protocol
- Standard Care Group (Active Comparator): Participants receive routine preoperative care according to standard clinical practice without ERAS-based nutrition education or fasting protocol.
  Interventions: Other: Standard Preoperative Care

INTERVENTIONS:
Behavioral: ERAS-Based Preoperative Nutrition Education and Fasting Protocol — A structured preoperative nutrition education program and evidence-based fasting protocol developed in accordance with ERAS guidelines, implemented during the 24 hours prior to total knee arthroplasty.
  Arms: ERAS-Based Preoperative Nutrition and Fasting Protocol Group
Other: Standard Preoperative Care — Participants receive routine preoperative care according to standard institutional clinical practice without ERAS-based nutrition education or fasting protocol.
  Arms: Standard Care Group

SUMMARY:
The aim of this randomized controlled study is to investigate the effect of implementing a preoperative nutrition education and fasting protocol prepared in accordance with Enhanced Recovery After Surgery (ERAS) guidelines during the 24-hour preoperative period on postoperative hydration status and the incidence of nausea and vomiting in patients scheduled for total knee arthroplasty.

Total knee arthroplasty is a commonly performed surgical procedure, particularly in older adults, and postoperative recovery may be negatively affected by surgical stress, anesthesia-related complications, dehydration, and postoperative nausea and vomiting. ERAS protocols emphasize the optimization of preoperative nutrition and hydration as key components to improve postoperative outcomes.

In this study, patients undergoing elective total knee arthroplasty will be randomly assigned to an intervention group or a control group. Patients in the intervention group will receive ERAS-based preoperative nutrition education and a standardized fasting protocol during the 24 hours prior to surgery, while patients in the control group will receive routine standard care.

Postoperative hydration status, nausea and vomiting severity, and fluid intake-output balance will be assessed and compared between the two groups. The findings of this study are expected to contribute to improving perioperative nursing care practices and enhancing patient recovery and comfort following total knee arthroplasty.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate the effect of ERAS protocol-based preoperative nutrition education and fasting management on postoperative hydration status and nausea-vomiting outcomes in patients undergoing elective total knee arthroplasty.

Total knee arthroplasty is an effective and frequently performed surgical intervention, particularly among older adults with degenerative joint disease. However, perioperative stress, prolonged fasting, and anesthesia-related factors may adversely affect postoperative recovery, leading to dehydration, nausea, and vomiting. Optimizing perioperative care through evidence-based ERAS protocols is therefore essential to improve patient outcomes.

ERAS protocols promote a multidisciplinary approach aimed at reducing surgical stress and accelerating postoperative recovery. One of the core components of ERAS is the optimization of preoperative nutrition and hydration. According to evidence-based guidelines, solid foods may be consumed up to 6 hours and clear liquids up to 2 hours prior to elective surgery. This approach reduces unnecessary prolonged fasting, prevents dehydration and insulin resistance, and improves postoperative comfort without increasing anesthesia-related risks.

The study will be conducted in the orthopedic clinic of Acıbadem Altunizade Hospital. Eligible patients scheduled for elective total knee arthroplasty will be recruited and randomly assigned to either the intervention or control group using a simple randomization method. Written informed consent will be obtained from all participants prior to enrollment.

Patients in the intervention group will receive an ERAS-based preoperative nutrition education leaflet and will be instructed to follow the standardized nutrition and fasting protocol during the 24-hour preoperative period. Patients in the control group will receive routine standard preoperative care as applied in the clinic.

Data collection will include demographic and clinical characteristics, postoperative hydration status, nausea and vomiting frequency and severity, and fluid intake-output monitoring. The following validated instruments will be used: the Surgical Thirst Discomfort Scale, the Rhodes Index of Nausea, Vomiting and Retching, a numeric nausea rating scale, and fluid balance monitoring forms.

Postoperative outcomes will be assessed for both groups, including hydration status, nausea and vomiting incidence, and fluid intake-output balance. Statistical analyses will be performed using SPSS software. Appropriate parametric or non-parametric tests will be applied based on data distribution, with a significance level set at p < 0.05.

This study aims to provide evidence on the effectiveness of ERAS-based preoperative nutrition education and fasting protocols in improving postoperative hydration and reducing nausea and vomiting, thereby supporting the development of structured, evidence-based nursing interventions in perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Adults aged 18 years and older.
* Patients scheduled for elective total knee arthroplasty.
* Patients expected to be hospitalized for at least 48 hours postoperatively.
* Ability to communicate verbally and provide informed consent.
* Patients with adequate cognitive and neurological capacity to understand study procedures.

Exclusion Criteria:

* Presence of any chronic disease requiring fluid restriction.
* Diagnosed cognitive impairment or psychiatric disorders affecting comprehension (e.g., Alzheimer's disease, dementia, psychotic disorders).
* Acute conditions causing dehydration in the preoperative period (e.g., vomiting, diarrhea, excessive fluid loss).
* Intraoperative complications requiring intensive care unit admission.
* Postoperative follow-up shorter than 48 hours due to early discharge or transfer to another clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Thirst Discomfort | Within the first 48 hours after surgery
  Postoperative thirst discomfort assessed using the Surgical Thirst Discomfort Scale. The scale includes 6 items (dry mouth, dry lips, thick saliva, dry throat, bad taste in the mouth, desire to drink water), each rated from 0 to 2 (0 = not uncomfortable, 1 = slightly uncomfortable, 2 = very uncomfortable). Total score range: 0-12. Higher scores indicate greater thirst-related discomfort (worse outcome).
Postoperative Fluid Balance | Within the first 48 hours after surgery
  Postoperative hydration status assessed by fluid intake-output balance records.

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting Severity | Within the first 48 hours after surgery
  Severity of postoperative nausea and vomiting assessed using the Rhodes Index of Nausea, Vomiting, and Retching (RINVR). The RINVR is an 8-item patient-reported scale. Each item is scored from 0 (no distress) to 4 (maximum distress), yielding a total score range of 0-32. Higher total scores indicate greater nausea/vomiting severity and distress (worse outcome).
Postoperative Nausea Intensity | Within the first 48 hours after surgery
  Intensity of postoperative nausea assessed using the Numeric Nausea Rating Scale (NNRS). Participants rate their current nausea severity on a numeric scale from 0 to 10, where 0 indicates no nausea and 10 indicates the most severe nausea. Higher scores indicate greater nausea intensity (worse outcome).
Perioperative Fluid Balance | From preoperative period to 48 hours postoperatively
  Perioperative fluid balance assessed as net fluid balance, calculated by subtracting total fluid output from total fluid intake using intake-output records.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Ocaktan, PhD, Principal Investigator — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acıbadem Health Group Atakent Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No